CLINICAL TRIAL: NCT00602979
Title: Prospective, Randomized Comparison of Intubating Conditions With Airtraq Optical, Storz DCI Video, McGRATH Video, GlideScope Video, & Macintosh Laryngoscope in Randomly Selected Elective Adult Surgical Patients
Brief Title: Comparison Study in Adult Surgical Patients of 5 Airway Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: King Systems Corporation (Industry); KARL STORZ Endoscopy-America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 0710009433
Record Dates: First submitted 2008-01-15; First posted 2008-01-28 (Estimated); Results first posted 2017-05-19 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2017-04

CONDITIONS: Laryngoscopy; Intubation
Keywords: endotracheal intubation; intubation; laryngoscopy; laryngoscope; surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- Macintosh laryngoscope (Other): Macintosh laryngoscope (control group/direct laryngoscopy) - current standard
  Interventions: Device: Macintosh laryngoscope
- Airtraq Optical Laryngoscope (Other): Airtraq® Optical Laryngoscope (an experimental group/indirect laryngoscopy)
  Interventions: Device: Airtraq® Optical Laryngoscope
- Storz DCI Video Laryngoscope (Other): Storz DCI Video Laryngoscope® (an experimental group/indirect laryngoscopy)
  Interventions: Device: Storz DCI Video Laryngoscope®
- GlideScope Video Laryngoscope (Other): GlideScope® Video Laryngoscope (an experimental group/indirect laryngoscopy)
  Interventions: Device: GlideScope® Video Laryngoscope
- McGRATH Video Laryngoscope (Other): McGRATH® Video Laryngoscope (an experimental group/indirect laryngoscopy)
  Interventions: Device: McGRATH® Video Laryngoscope

INTERVENTIONS:
Device: Macintosh laryngoscope — Used during laryngoscopy to facilitate intubation.
  Arms: Macintosh laryngoscope
Device: Airtraq® Optical Laryngoscope — Used during laryngoscopy to facilitate intubation.
  Arms: Airtraq Optical Laryngoscope
Device: Storz DCI Video Laryngoscope® — Used during laryngoscopy to facilitate intubation
  Arms: Storz DCI Video Laryngoscope
Device: GlideScope® Video Laryngoscope — Used during laryngoscopy to facilitate intubation
  Arms: GlideScope Video Laryngoscope
Device: McGRATH® Video Laryngoscope — Used during laryngoscopy to facilitate intubation
  Arms: McGRATH Video Laryngoscope

SUMMARY:
The placement of endotracheal tubes (intubation) is a physiologically stressful procedure for patients. Laryngoscopes are devices-typically composed of a blade attached to a handle with a light source-that allow examination of the upper airway through the mouth, often for the purposes of intubation. Recently some new laryngoscope devices (including the Airtraq® Optical Laryngoscope, the Storz DCI Video laryngoscope®, McGRATH® Video Laryngoscope, and the GlideScope®) have been developed, which may either decrease the stress related to intubation (reduce neck extension, reduce risk of complications or reduce time elapsed during intubation) or improve intubation success (reduce the number of attempts at intubating). Data are being collected in this study to determine which of these commonly-used devices may be better, particularly in comparison to the current hospital standard, the Macintosh laryngoscope. All of the devices to be used in this study are currently cleared or exempt by the Food and Drug Administration (FDA).

DETAILED DESCRIPTION:
Historically, optical and video laryngoscopes have been used as alternative airway management devices for the difficult airway, and as rescue devices. Their use by experienced laryngoscopists has not been compared in a prospective, randomized, head-to-head comparison for routine airway management in adult surgical patients. Video and optical laryngoscopes have been developed to improve the laryngeal view for tracheal intubation and to decrease physiological stress associated with the procedure. The objective of this study is to determine whether these devices offer superior intubating conditions for routine surgical management, over the Macintosh laryngoscope, which is the current standard. The devices to be compared in this study are the most commonly used video and optical laryngoscopes on the market and are cleared or exempt by the Food and Drug Administration (FDA).

Eligible subjects include elective adult surgical patients with an ASA status between 1 and 3 requiring general endotracheal anesthesia. Subjects with a BMI ≥ 40, or undergoing surgery in close proximity to the neck will be excluded. Prior to surgery, subjects will receive a pre-anesthesia evaluation with particular attention to the airway using the Mallampati classification system; atlanto-occipital joint extension; thyro-mental distance; temporomandibular joint function; inter-incisor distance; and dental assessment. Subjects will be randomized for intubation with one of the five laryngoscopes in equal proportions. The following data were recorded: total intubation time, maximum neck extension using an angle gauge, glottic view, assessed by the anesthesiologist using the Cook modification of the Cormack-Lehane grading system (Figure 1), and ease of tracheal intubation using a 5-point rating scale; 5 (excellent) to 1 (poor). Subjects were queried about soreness or painful swallowing in the PACU and a week later via a phone call.

ELIGIBILITY:
Inclusion Criteria:

* Elective adult surgical patient requiring general endotracheal anesthesia.
* Males and Females.
* ASA Physical Status 1-3.
* Age 18 years of age and older

Exclusion Criteria:

* Body Mass Index (BMI) ≥35kg/m2.
* If subject is of childbearing potential, a positive pregnancy test at the time of study enrollment.
* Has physical, mental, or medical conditions which, in the opinion of the Investigator, could compromise the subject's welfare, ability to communicate with the study staff, complete study activities, or would otherwise contraindicate study participation.
* Intubated prior to surgery.
* Severe cardiovascular, hepatic or renal disease.
* Need for nasal intubation.
* An investigator of this study.
* Inclusion in another clinical research study.
* Subject's refusal or inability to agree to and to sign the Informed Consent Form in English.
* Subject requiring awake airway management.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2008-04; Primary Completion 2009-09 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon Samuels, MD, Principal Investigator — Weill Medical College of Cornell University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cook TM. A new practical classification of laryngeal view. Anaesthesia. 2000 Mar;55(3):274-9. doi: 10.1046/j.1365-2044.2000.01270.x. PMID 10671848

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Macintosh Laryngoscope | Airtraq Optical Laryngoscope | Storz DCI Video Laryngoscope | GlideScope Video Laryngoscope | McGRATH Video Laryngoscope
Started | 48 | 48 | 48 | 48 | 48
Completed | 45 | 45 | 45 | 45 | 45
Not Completed | 3 | 3 | 3 | 3 | 3
Not completed — Lost to Follow-up | 3 | 2 | 3 | 2 | 3
Not completed — Failed Intubation | 0 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Macintosh Laryngoscope | Airtraq Optical Laryngoscope | Storz DCI Video Laryngoscope | GlideScope Video Laryngoscope | McGRATH Video Laryngoscope | Total
Number analyzed (Participants) | 48 | 48 | 48 | 48 | 48 | 240
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (16.9) | 46.1 (13.5) | 47.8 (15.4) | 50.0 (15.2) | 49.3 (15.8) | 48.7 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 25 | 21 | 25 | 23 | 114
  Male | 28 | 23 | 27 | 23 | 25 | 126

OUTCOME MEASURES:

1. Primary Outcome: Percentage Distribution of Cook's Modification of Cormack-Lehane's Grading System. Each Study Subject Will Receive a Grade of 1, 2A, 2B, 3A, 3B, or 4 in the Cormack-Lehane Grading System.
Description: Percentage distribution of Cook's modification of Cormack-Lehane's grading system. This is a classification that records the best laryngeal view obtained with or without anterior laryngeal pressure. Each study subject will receive a grade of 1, 2A, 2B, 3A, 3B, or 4 in the Cormack-Lehane grading system. Grades 1 and 2A classify as an easy view: when the laryngeal inlet is visible. Grades 2B and 3A classify as restricted: when the posterior glottic structures are visible or the epiglottis is visible and can be lifted. Grades 3B and 4 classify as difficult: when the epiglottis cannot be lifted or when no laryngeal structures are visible.
  Cook's modification of Cormack-Lehane's Grades 1=1, 2=2A,3=2B, 4=3A, 5=3B, 6=4.
Time Frame: 1 time during laryngoscopy
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Macintosh Laryngoscope | Airtraq Optical Laryngoscope | Storz DCI Video Laryngoscope | GlideScope Video Laryngoscope | McGRATH Video Laryngoscope
Number analyzed (Participants) | 45 | 45 | 45 | 45 | 45
units on a scale | 1.98 (1.96) | 1.18 (0.44) | 1.27 (0.54) | 1.47 (0.59) | 1.13 (0.34)

ADVERSE EVENTS:
Arm/Group | Macintosh Laryngoscope | Airtraq Optical Laryngoscope | Storz DCI Video Laryngoscope | GlideScope Video Laryngoscope | McGRATH Video Laryngoscope
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/48 | 0/48 | 0/48 | 0/48
Serious Adverse Events (participants affected / at risk) | 2/48 | 0/48 | 0/48 | 0/48 | 1/48
Other Adverse Events (participants affected / at risk) | 0/48 | 0/48 | 0/48 | 0/48 | 1/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Macintosh Laryngoscope (N=48) | Airtraq Optical Laryngoscope (N=48) | Storz DCI Video Laryngoscope (N=48) | GlideScope Video Laryngoscope (N=48) | McGRATH Video Laryngoscope (N=48)
Corneal Laceration (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iliac Vein Rupture (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Right Tonsillar Pillar Laceration (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Macintosh Laryngoscope (N=48) | Airtraq Optical Laryngoscope (N=48) | Storz DCI Video Laryngoscope (N=48) | GlideScope Video Laryngoscope (N=48) | McGRATH Video Laryngoscope (N=48)
Swollen Lip (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No